CLINICAL TRIAL: NCT05902832
Title: Computer-Mediated Intervention to Enhance Emotional Competence in Children With Autism in Schools
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Ofer Golan, Prof. Ofer Golan, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Bar Ilan University
Record Dates: First submitted 2023-02-09; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability, Mild
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: participant will be randomly divided to one of two groups: first group will take part in the intervention program and the second will be wait-listed and children will receive treatment as usual
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group - Autistic children (Experimental): 60 7-10-years-old autistic children, from special education classes integrated in regular schools.
  this group will receive EmotiPlay's intervention in the curriculum.
  Interventions: Behavioral: EmotiPlay
- Control group- Autistic children (No Intervention): 60 7-10-years-old autistic children, from special education classes integrated in regular schools.
  this group will be wait-listed and receive treatment as usual.
- Control group-Neurotypical (No Intervention): 30 6-10-years-old children, from regular education match in cognitive and linguistic abilities.

INTERVENTIONS:
Behavioral: EmotiPlay — EmotiPlay is a computer-based intervention program, designed to enhance emotion recognition (ER) by addressing multiple modalities of emotional cues (facial expressions, tone of voice, body language),
  Arms: Experimental group - Autistic children

SUMMARY:
Autism spectrum condition (ASC) is a neurodevelopmental disorder characterized fundamentally by social deficits. Emotional competence - the ability to express, recognize, understand, and regulate emotions - is a key aspect of social communication. Evidence suggests that the developmental trajectories of autistic children differ from that of neuro-typical children regarding their ability to process and recognize emotions from paralinguistic emotional facial, body language, and voice tone cues. They also have difficulty integrating these cues in context and lack in emotional language.

Numerous approaches to teaching people with autism how to recognize and understand emotions have been tried, with recent increased interest in computer-based interventions (CBI). However, most of the research focused only on facial expressions, were limited to autistic children with no intellectual disabilities (ID); and showed limited generalization to real social settings. EmotiPlay, a computer-based intervention program, designed to enhance emotion recognition (ER) by addressing multiple modalities of emotional cues (facial expressions, tone of voice, body language), has shown good outcome when used at home by autistic children and no ID . However, the examination of generalization was partial and depended only on parental reports.

The present study main goals are to: (1) Examine the adaptation and the integration of EmotiPlay into special education classrooms in regular schools. (2) Assess EmotiPlay's effect on emotional competence among autistic children at different functioning levels.

DETAILED DESCRIPTION:
This research is comprised of two main stages:

the first stage is a Pilot, who's main goals are to examine the adaptation and integration of EmotiPlay's intervention to a school setting with autistic children at various ages and levels of functioning, and to test an extended EC battery for EmotiPlay's evaluation.

The pilot includes 5 special education classes that will take part at a short version of the intervention program, and a control group of neurotypical children matched in intellectual and linguistic abilities.

the second stage will include 150 participants, divided into three groups: 60 7-10-year-old autistic children who will participate in the intervention program; 60 7-10-year-old autistic children who will not participate in the intervention; and 30 neuro-typical children matched in cognitive and linguistic skills.

All participant will undergo a pre-assessment tests that include: (1) multi-modal basic and complex ER (2) emotion understanding based on a standardized measure (the Test of Emotion Comprehension - TEC) (3) an emotion definition task (4) a story- telling task (5) an observation of children's prosocial behavior during free-playtime (using the Playground Observation of Peer Engagement - POPE). After evaluations participants will be randomly divided into two groups, the first group will take part in the intervention program and the second will be the control group.

EmotiPlay's intervention program will be administered by a certified educational staff for 18 weeks (36 lessons).

All participant will be evaluated immediately after the intervention; and 15 weeks post-intervention.

The important contribution of this study is twofold. It integrates an intervention program to promote emotional competence into the educational system, which serves as a major platform for acquiring social skills. Concurrently, it offers a way to assess the social functioning in real life situations of children with autism at different levels of functioning.

ELIGIBILITY:
Inclusion Criteria:

* autism spectrum condition

Exclusion Criteria:

* Verbal Intelligence (according to Wechsler) 3 or lower.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Emotion recognition task | before intervention
  Emotion recognition test includes 4 tasks to examine emotion recognition: 1. facial expressions videos 2. decontextualized vocal utterances 3. body language videos 4. Integrative video clips presenting all 3 modalities in context, that were extracted from old television shows, sound track was muffled in order to prevent semantic information, but keep prosodic cues. The test include 12 emotions, for every video or recording 4 answers are presented, the target emotion and the order of the possible answers was counterbalanced. In each modality the subject can achieve 0-12 points, a point for every emotion recognized correctly.
Emotion recognition | immediately after the intervention
  Emotion recognition test includes 4 tasks to examine emotion recognition: 1. facial expressions videos 2. decontextualized vocal utterances 3. body language videos 4. Integrative video clips presenting all 3 modalities in context, that were extracted from old television shows, sound track was muffled in order to prevent semantic information, but keep prosodic cues. The test include 12 emotions, for every video or recording 4 answers are presented, the target emotion and the order of the possible answers was counterbalanced. In each modality the subject can achieve 0-12 points, a point for every emotion recognized correctly.
Emotion recognition | 15 weeks after the end of the intervention
  Emotion recognition test includes 4 tasks to examine emotion recognition: 1. facial expressions videos 2. decontextualized vocal utterances 3. body language videos 4. Integrative video clips presenting all 3 modalities in context, that were extracted from old television shows, sound track was muffled in order to prevent semantic information, but keep prosodic cues. The test include 12 emotions, for every video or recording 4 answers are presented, the target emotion and the order of the possible answers was counterbalanced. In each modality the subject can achieve 0-12 points, a point for every emotion recognized correctly.
Emotion understanding | before intervention
  TEC - Test of Emotion Competence (Pons & Harris, 2000) design to assess emotion understanding in 3-12 years old children, it is based on Pons et al. (2002) model of 9 developmental stages to emotion understanding among children.
  In the test, the subjects are presented with 23 illustrated pictures, in a boy and girl versions. In the first 5 scenarios the child is asked to recognize basic emotions from facial expressions, Next, the child is presented with short stories and the illustrated picture is missing emotional cues in the character face. The examiner reads the story and the child is asked to choose the correct emotion from 4 options. Maximum scoring 21 points.
Emotion understanding | immediately after the intervention
  TEC - Test of Emotion Competence (Pons & Harris, 2000) design to assess emotion understanding in 3-12 years old children, it is based on Pons et al. (2002) model of 9 developmental stages to emotion understanding among children.
  In the test, the subjects are presented with 23 illustrated pictures, in a boy and girl versions. In the first 5 scenarios the child is asked to recognize basic emotions from facial expressions, Next, the child is presented with short stories and the illustrated picture is missing emotional cues in the character face. The examiner reads the story and the child is asked to choose the correct emotion from 4 options. Maximum scoring 21 points.
Emotion understanding | 15 weeks after the end of the intervention
  TEC - Test of Emotion Competence (Pons & Harris, 2000) design to assess emotion understanding in 3-12 years old children, it is based on Pons et al. (2002) model of 9 developmental stages to emotion understanding among children.
  In the test, the subjects are presented with 23 illustrated pictures, in a boy and girl versions. In the first 5 scenarios the child is asked to recognize basic emotions from facial expressions, Next, the child is presented with short stories and the illustrated picture is missing emotional cues in the character face. The examiner reads the story and the child is asked to choose the correct emotion from 4 options. Maximum scoring 21 points.
Emotional-mental vocabulary | before intervention
  Emotion definition task - assess the subject's ability to define 12 emotions. Participants were asked to define the emotion (for example: "please explain what is happy?") and to give examples to personalize experience related to each of the emotions (e.g.: "can you describe a situation that you felt happy?"). The definition and examples were audiotaped, and then transcribed. Points will be allocated to the definition of each emotion according the subscale vocabulary in WISC- IV, all emotions falls within the range of 0 to 24 points
Emotional-mental vocabulary | immediately after the intervention
  Emotion definition task - assess the subject's ability to define 12 emotions. Participants were asked to define the emotion (for example: "please explain what is happy?") and to give examples to personalize experience related to each of the emotions (e.g.: "can you describe a situation that you felt happy?"). The definition and examples were audiotaped, and then transcribed. Points will be allocated to the definition of each emotion according the subscale vocabulary in WISC- IV, all emotions falls within the range of 0 to 24 points
Emotional-mental vocabulary | 15 weeks after the end of the intervention
  Emotion definition task - assess the subject's ability to define 12 emotions. Participants were asked to define the emotion (for example: "please explain what is happy?") and to give examples to personalize experience related to each of the emotions (e.g.: "can you describe a situation that you felt happy?"). The definition and examples were audiotaped, and then transcribed. Points will be allocated to the definition of each emotion according the subscale vocabulary in WISC- IV, all emotions falls within the range of 0 to 24 points
social functioning | before intervention
  socio-emotional functioning will be evaluated by playground observation and coded by POPE - Playground Observation of Peer Engagement (Kasari et al, 2005). This instrument is a time-interval behavior coding system. Independent observers from the research team watched the target child on the playground for 40 consecutive seconds and then coded for 2 seconds for ten minutes during school recess. The observers noted the child's engagement with peers on the playground (solitary, proximity, onlooking, parallel, parallel aware, involved in games and rules and joint engaged with peers) in each interval. Coders will also note positive and negative initiations of the target child towered other children, and positive and negative responses to a peer's social overtures.
social functioning | immediately after the intervention
  socio-emotional functioning will be evaluated by playground observation and coded by POPE - Playground Observation of Peer Engagement (Kasari et al, 2005). This instrument is a time-interval behavior coding system. Independent observers from the research team watched the target child on the playground for 40 consecutive seconds and then coded for 2 seconds for ten minutes during school recess. The observers noted the child's engagement with peers on the playground (solitary, proximity, onlooking, parallel, parallel aware, involved in games and rules and joint engaged with peers) in each interval. Coders will also note positive and negative initiations of the target child towered other children, and positive and negative responses to a peer's social overtures.
social functioning | 15 weeks after the end of the intervention
  socio-emotional functioning will be evaluated by playground observation and coded by POPE - Playground Observation of Peer Engagement (Kasari et al, 2005). This instrument is a time-interval behavior coding system. Independent observers from the research team watched the target child on the playground for 40 consecutive seconds and then coded for 2 seconds for ten minutes during school recess. The observers noted the child's engagement with peers on the playground (solitary, proximity, onlooking, parallel, parallel aware, involved in games and rules and joint engaged with peers) in each interval. Coders will also note positive and negative initiations of the target child towered other children, and positive and negative responses to a peer's social overtures.
spontaneous emotional mental language | before intervention
  Narrative re-telling task - narratives were elicited using two wordless picture-books, "Frog on His Own (Mayer, 1973) and "Frog, where are you?" (Mayer, 1969). Stories were shortened to a 15-pages, depicting a frog's adventures after departing from his boy companion. Participants are asked to listen to a story the examiner is telling with a predetermined script, while presenting the pictures on an iPad (via book creator app). One book was randomly assigned to each participant, and after listening to the story, the participants will be asked to tell the story in their own words while flipping through the pictures.
  The stories will be audiotaped, transcribed and coded according to Capps et al., (2000)
spontaneous emotional mental language | immediately after the intervention
  Narrative re-telling task - narratives were elicited using two wordless picture-books, "Frog on His Own (Mayer, 1973) and "Frog, where are you?" (Mayer, 1969). Stories were shortened to a 15-pages, depicting a frog's adventures after departing from his boy companion. Participants are asked to listen to a story the examiner is telling with a predetermined script, while presenting the pictures on an iPad (via book creator app). One book was randomly assigned to each participant, and after listening to the story, the participants will be asked to tell the story in their own words while flipping through the pictures.
  The stories will be audiotaped, transcribed and coded according to Capps et al., (2000)
spontaneous emotional mental language | 15 weeks after the end of the intervention
  Narrative re-telling task - narratives were elicited using two wordless picture-books, "Frog on His Own (Mayer, 1973) and "Frog, where are you?" (Mayer, 1969). Stories were shortened to a 15-pages, depicting a frog's adventures after departing from his boy companion. Participants are asked to listen to a story the examiner is telling with a predetermined script, while presenting the pictures on an iPad (via book creator app). One book was randomly assigned to each participant, and after listening to the story, the participants will be asked to tell the story in their own words while flipping through the pictures.
  The stories will be audiotaped, transcribed and coded according to Capps et al., (2000)

SECONDARY OUTCOMES:
Autistic traits | before the intervention
  The school-age form (4 to 18 years) of the Social Responsiveness Scale, 2nd edition (SRS-2) (Constantino & Gruber, 2012) to assess severity of autism traits.
  The SRS-2 measures social awareness, social communication, social motivation, social cognition and inflexible behaviors applying a dimensional concept of autism. The SRS-2 includes 65 items., each scored on a 4-point Likert scale, from 0 ("not true") to 3 ("almost always true"), yielding a maximum of 195. Out of the 65 items of the SRS-2, 53 focus on social communicative abilities, these items examine the ability to interpret social cues, to maintain social conversation, as well as to initiate social interaction (e.g., "Doesn't recognize when others are trying to take advantage of him or her"). The 12 remaining items probe repetitive behaviors or restricted patterns of interest (e.g., "Shows unusual sensory interests or strange ways of playing with toys").
Autistic traits | immediately after the intervention
  The school-age form (4 to 18 years) of the Social Responsiveness Scale, 2nd edition (SRS-2) (Constantino & Gruber, 2012) to assess severity of autism traits.
  The SRS-2 measures social awareness, social communication, social motivation, social cognition and inflexible behaviors applying a dimensional concept of autism. The SRS-2 includes 65 items., each scored on a 4-point Likert scale, from 0 ("not true") to 3 ("almost always true"), yielding a maximum of 195. Out of the 65 items of the SRS-2, 53 focus on social communicative abilities, these items examine the ability to interpret social cues, to maintain social conversation, as well as to initiate social interaction (e.g., "Doesn't recognize when others are trying to take advantage of him or her"). The 12 remaining items probe repetitive behaviors or restricted patterns of interest (e.g., "Shows unusual sensory interests or strange ways of playing with toys").
adaptive skills | before the intervention
  ABAS-II: Adaptive Behavior Assessment System (Harrison & Oakland, 2003), assessment of the adaptive skills of individuals. This measure evaluates 10 adaptive domains: communication. Functional academics, self-direction. Leisure, social. Community use, home / school living health and safety, self-care and work. ABAS-II was translated to Hebrew and standardized by PsychTech Ltd.
adaptive skills | immediately after the intervention
  ABAS-II: Adaptive Behavior Assessment System (Harrison & Oakland, 2003), assessment of the adaptive skills of individuals. This measure evaluates 10 adaptive domains: communication. Functional academics, self-direction. Leisure, social. Community use, home / school living health and safety, self-care and work. ABAS-II was translated to Hebrew and standardized by PsychTech Ltd.

CONTACTS AND LOCATIONS:
Locations (1):
- Bar Ilan University, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fridenson-Hayo S, Berggren S, Lassalle A, Tal S, Pigat D, Bolte S, Baron-Cohen S, Golan O. Basic and complex emotion recognition in children with autism: cross-cultural findings. Mol Autism. 2016 Dec 19;7:52. doi: 10.1186/s13229-016-0113-9. eCollection 2016. PMID 28018573
- [Result] Golan O, Baron-Cohen S, Golan Y. The 'Reading the Mind in Films' Task [child version]: complex emotion and mental state recognition in children with and without autism spectrum conditions. J Autism Dev Disord. 2008 Sep;38(8):1534-41. doi: 10.1007/s10803-007-0533-7. Epub 2008 Feb 29. PMID 18311514
- [Result] Macrostructure, microstructure, and mental state terms in the narratives of English-Hebrew bilingual preschool children with and without specific language impairment. Applied PsychoLinguistics, 37(1), 165-193.